CLINICAL TRIAL: NCT07128706
Title: Harmonization and Implementation of Sports-related Concussion Guidelines in European Football for Youth - the REFORM Erasmus + Project
Brief Title: Harmonization and Implementation of Sports-related Concussion Guidelines in European Football for Youth - the Erasmus + Project
Acronym: REFORM
Status: Enrolling by invitation | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Universität des Saarlandes (Other); UiT The Arctic University of Norway (Other); University Hospital of Split (Other)
Responsible Party: Sponsor
Other Study IDs: 101133951
Record Dates: First submitted 2025-07-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Sports-related Concussion
Keywords: awareness; european football; youth; sports-related concussions; management; education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study addresses the evident gap in SRC awareness and reporting, especially at the grassroots level, by harmonizing concussion management practices across Europe and observing its impact on stakeholders' (coaches, parents, players, referees) knowledge and practices.

DETAILED DESCRIPTION:
This project is a multi-phase observational study using a participatory action research design. It includes the identification, documentation, and evaluation of educational tools to improve concussion management practices in European youth football. Each phase of the study is guided by the Logical Framework Approach (LFA) to ensure systematic evaluation and measurable outcomes.

The project adopts a stakeholder-centered methodology, involving key stakeholders, including football associations, healthcare professionals, and academia, from Norway, Germany, Croatia, and Türkiye. This structured approach ensures that each phase aligns with specific objectives, outputs, and outcomes, enhancing the project's coherence and impact. The LFA was chosen for its structured, outcome-oriented methodology, which aligns well with the goals of this multi-phase, transnational project. LFA facilitates clear goal-setting, stakeholder engagement, and systematic monitoring, ensuring alignment between the project's objectives and measurable outcomes. Compared to other participatory research approaches, LFA's emphasis on stakeholder-driven planning ensures that the developed educational tools are practical, culturally relevant, and widely applicable across diverse European football contexts.

The project will use a stakeholder approach to collaboratively observe, assess, and document innovative educational materials and resources for concussion awareness that emerging in routine practice. This process will be interdisciplinary and transnational, ensuring that the materials are harmonized and build upon each other to meet the needs of various stakeholders. The project will use surveys to articulate training and educational standards to ensure a high-quality standard that can be scaled across European national football associations down to grassroots levels in each country.

Through a participatory process, the project will solicit expert opinion and keep an ongoing dialogue with multiple facets of stakeholders to guarantee an evidence-based joint European educational awareness set that meets the demands of the coaches and board, as well as fostering an awareness in the players and their families.

Setting and Participants The project will be conducted in collaboration with football associations from Norway, Germany, Croatia, and Türkiye. Participants will include selected football clubs from these countries, chosen to represent diverse cultural and operational contexts.

To ensure the educational materials are effective across the diverse cultural contexts of the participating countries, the project will implement a robust process of cultural adaptation. This will involve the translation of educational materials into the native languages of each participating country, ensuring accuracy and clarity in communication. UEFA-approved translators will be used to maintain the integrity of the content.

Additionally, local experts, football stakeholders, and national football federations will play an active role in providing culturally specific insights throughout the development phase. This collaborative approach ensures that the content resonates with the distinct cultural contexts, communication styles, and practices of each country. Focus group discussions and pilot testing will be conducted in each country to refine the materials further, ensuring their relevance and effectiveness in addressing regional nuances related to concussion management.

The dissemination phase employs a multi-channel strategy, combining direct stakeholder engagement with digital tools and institutional partnerships to reach diverse audiences across Europe. Resources will be shared with national football associations for scaling across Europe, leveraging social media platforms to enhance outreach. The findings of this project will be analyzed and published in peer-reviewed journals, as well as presented at key conferences. All findings will be disseminated to accurately inform future practices. This will occur immediately after the completion of the final analysis.

ELIGIBILITY:
Inclusion Criteria:

Clubs: Youth football clubs in the four countries will be invited to participate. Clubs must have:

* The ability to implement new concussion protocols with support from the project team. This will include basic resources such as access to digital platforms (e.g., internet connectivity, devices to access training materials).
* A willingness to engage with and integrate educational materials into their regular operations. Federations will support clubs in understanding these expectations before participation.

Stakeholders: Key stakeholder groups involved in youth football will be included:

* Coaches of youth teams, regardless of prior experience in concussion management.
* Players actively participating in youth football (targeting diverse age groups and genders).
* Parents of youth players to ensure comprehensive inclusion of perspectives.
* Referees involved in officiating youth football matches.
* Medical personnel, including team doctors and physiotherapists.

Exclusion Criteria:

* Clubs that lack the basic resources or logistical capacity to access digital learning platforms or implement concussion protocols (as determined by federations).
* Stakeholders who are unwilling to participate or unable to provide informed consent (or, for minors, parental/guardian consent).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Coaches, referees, parents and youth football players (up to U23) involved in football federations among Croatia, Norway, Germany and Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Concussion Knowledge Score Pre- and Post-Educational Toolkit | Baseline (pre-intervention) and up to 4 weeks post-intervention
  Concussion knowledge will be assessed using a structured multiple-choice questionnaire developed for this study, based on international concussion education guidelines. The same test will be administered immediately before the educational intervention (toolkit) and within 4 weeks after completion. Each correct answer is scored as 1 point. The total score ranges from 0 to 25. Higher scores indicate greater knowledge.

SECONDARY OUTCOMES:
Number of Participants Completing the Online Concussion Education Course (MOOC) | Within 6 weeks after enrollment in the course
  Engagement with the online concussion education course will be measured by tracking completion data through the course platform. Completion is defined as finishing all mandatory modules and quizzes. Data will be automatically recorded and exported from the course analytics dashboard.
Number of Clubs Utilizing the Educational Toolkit | Up to 3 months after intervention rollout
  Toolkit utilization will be assessed via club reports and checklists submitted at the end of the intervention period. Clubs will indicate which toolkit components (e.g., posters, handouts, team briefings) were used. A club is considered a user if at least one core component was implemented.
Number of Participants Attending Live Concussion Education Workshops | Throughout the intervention period (approx. 3 months)
  Attendance at live in-person or virtual workshops will be tracked through registration lists and sign-in sheets. Workshop participation will be considered complete if the participant attended at least 80% of the session.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
data are anonymously collected